CLINICAL TRIAL: NCT01409577
Title: Clinical Outcome of Fractional Flow Reserve-guided Coronary Intervention Strategy in Koreans
Brief Title: Outcome of FFR-guided Intervention Strategy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Collaborators: Ajou University (Other); Keimyung University Dongsan Medical Center (Other); Inje University (Other)
Responsible Party: Principal Investigator, Bon-Kwon Koo, Associate professor, Seoul National University Hospital
Other Study IDs: H1102-032-350
Record Dates: First submitted 2011-08-02; First posted 2011-08-04 (Estimated); Last update posted 2011-11-22 (Estimated); Status verified 2011-11

CONDITIONS: Coronary Artery Disease
Keywords: Coronary stenosis; stent; fractional flow reserve
MeSH Terms: conditions — Coronary Artery Disease; Coronary Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- FFR: Patients with intermediate coronary stenosis Patients with successful fractional flow measurement Feasible > 9months clinical follow-up

SUMMARY:
The investigator will evaluate the clinical outcomes of the patients in whom the treatment strategy for their coronary stenosis were determined by fractional flow reserve measurement.

DETAILED DESCRIPTION:
Inclusion criteria

* Coronary stenosis
* Successful measurement of fractional flow reserve

Clinical outcomes

* Death
* Cardiac death
* Target lesion revascularization
* Target vessel revascularization

ELIGIBILITY:
Inclusion Criteria:

* Coronary stenosis
* Successful fractional flow reserve measurement

Exclusion Criteria:

* Contraindication to adenosine
* Expected life expectance < 1year

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with intermediate coronary stenosis by visual estimation
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2011-03; Primary Completion 2011-12 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
Long-term MACE | 5 years
  Cardiac death, MI, target vessel revascularization, target lesion revascularization

SECONDARY OUTCOMES:
Short-term MACE | 9 months
  Cardiac death, MI, TLR/TVR

CONTACTS AND LOCATIONS:
Overall Officials: Bon-Kwon Koo, MD, PhD, Principal Investigator — Seoul National University
Locations (2):
- South Korea (2):
  - Ilsan Paik hospital, Ilsan
  - Seoul National University Hospital, Seoul